CLINICAL TRIAL: NCT02013687
Title: A Phase 1 Study of the Safety and Immunogenicity of Plant-Derived Pfs25 VLP-FhCMB Malaria Transmission Blocking Vaccine in Healthy Adults
Brief Title: Safety and Immunogenicity of Plant-Derived Pfs25 VLP-FhCMB Malaria Transmission Blocking Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fraunhofer, Center for Molecular Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FhCMB Pfs25-001
Record Dates: First submitted 2013-11-25; First posted 2013-12-17 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 2 µg + Alhydrogel (Experimental): vaccine
  Interventions: Biological: Pfs25 VLP- FhCMB
- 10 µg + Alhydrogel (Experimental): vaccine
  Interventions: Biological: Pfs25 VLP- FhCMB
- 30 µg + Alhydrogel (Experimental): vaccine
  Interventions: Biological: Pfs25 VLP- FhCMB
- 100 µg + Alhydrogel (Experimental): vaccine
  Interventions: Biological: Pfs25 VLP- FhCMB

INTERVENTIONS:
Biological: Pfs25 VLP- FhCMB

SUMMARY:
This study is a Phase 1, dose escalation, first-in-human study designed primarily to evaluate the safety of the purified plant-derived Pfs25 VLP combined with Alhydrogel adjuvant

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female aged 18 - 50 years inclusive
* Able to give written informed consent obtained prior to screening
* Healthy, as determined by medical history, physical examination, vital signs, and clinical safety laboratory examinations at baseline
* Women of childbearing potential must have a negative urine pregnancy test within 24 hours preceding receipt of each dose.
* Females should fulfill one of the following criteria:

  1. At least one year post-menopausal
  2. Surgically sterile
  3. Willing to use oral, implantable, transdermal or injectable contraceptives for 30 days prior to first vaccination and then for the study duration
  4. Willing to abstain from sexual intercourse or use another reliable form of contraception approved by the Investigator (e.g., intrauterine device (IUD), female condom, diaphragm with spermicide, cervical cap, use of condom by the sexual partner or a sterile sexual partner) for 30 days prior to first vaccination through 9 months after third vaccination
* Comprehension of the study requirements, as demonstrated by achieving a score of at least 80% correct on a short multiple-choice quiz.

  * Individuals who fail to achieve a passing score on the initial comprehension assessment will be given the opportunity to retest after a review of protocol information.
  * Individuals who fail the comprehension assessment for the second time will not be enrolled.
* Available and able to participate in all planned study visits and procedures.

Exclusion Criteria:

* History of malaria or previous receipt of an investigational malaria vaccine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Accelovance, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chichester JA, Green BJ, Jones RM, Shoji Y, Miura K, Long CA, Lee CK, Ockenhouse CF, Morin MJ, Streatfield SJ, Yusibov V. Safety and immunogenicity of a plant-produced Pfs25 virus-like particle as a transmission blocking vaccine against malaria: A Phase 1 dose-escalation study in healthy adults. Vaccine. 2018 Sep 18;36(39):5865-5871. doi: 10.1016/j.vaccine.2018.08.033. Epub 2018 Aug 17. PMID 30126674

RESULTS

PARTICIPANT FLOW:
Groups:
- 2 µg + Alhydrogel; 10 µg + Alhydrogel; 30 µg + Alhydrogel; 100 µg + Alhydrogel: Pfs25 VLP- FhCMB vaccine
Period: Overall Study
Arm/Group | 2 µg + Alhydrogel | 10 µg + Alhydrogel | 30 µg + Alhydrogel | 100 µg + Alhydrogel
Started | 6 | 6 | 16 | 16
Completed | 6 | 6 | 14 | 14
Not Completed | 0 | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Missed visits due to patient travel | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 µg + Alhydrogel | 10 µg + Alhydrogel | 30 µg + Alhydrogel | 100 µg + Alhydrogel | Total
Number analyzed (Participants) | 6 | 6 | 16 | 16 | 44
Age, Customized [Mean (Standard Deviation); unit: years] | 36.8 (8.93) | 36.7 (6.59) | 36.1 (8.96) | 30.6 (8.86) | 34.3 (8.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 7 | 5 | 18
  Male | 3 | 3 | 9 | 11 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 1 | 5
  Not Hispanic or Latino | 4 | 5 | 15 | 14 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 10 | 11 | 28
  White | 2 | 2 | 6 | 5 | 15
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Subjects With at Least One Adverse Event
Time Frame: 336 days
Measure: Count of Participants; unit: Participants
Arm/Group | 2 µg + Alhydrogel | 10 µg + Alhydrogel | 30 µg + Alhydrogel | 100 µg + Alhydrogel
Number analyzed (Participants) | 6 | 6 | 16 | 16
Participants | 4 | 4 | 11 | 15

2. Primary Outcome: Subjects With Solicited Systemic Adverse Events
Time Frame: 336 days
Measure: Count of Participants; unit: Participants
Groups:
- 2 µg + Alhydrogel; 10 µg + Alhydrogel; 30 µg + Alhydrogel; 100 µg + Alhydrogel: Pfs25 VLP-FhCMB vaccine
Arm/Group | 2 µg + Alhydrogel | 10 µg + Alhydrogel | 30 µg + Alhydrogel | 100 µg + Alhydrogel
Number analyzed (Participants) | 6 | 6 | 16 | 16
Participants | 2 | 4 | 8 | 10

3. Primary Outcome: Subjects With Solicited Local Adverse Events
Time Frame: 336 days
Measure: Count of Participants; unit: Participants
Arm/Group | 2 µg + Alhydrogel | 10 µg + Alhydrogel | 30 µg + Alhydrogel | 100 µg + Alhydrogel
Number analyzed (Participants) | 6 | 6 | 16 | 16
Participants | 4 | 6 | 12 | 15

4. Secondary Outcome: Assessment of Anti-Pfs25 IgG Following the Third Immunization.
Description: Serum anti-Pfs25 antibody IgG titers determined using an ELISA unit assay.
Time Frame: 196 days
Population: In the "30 µg + Alhydrogel" group, 15 out of 16 patient samples were analyzed as 1 patient in the group had withdrawn from the study by study day 196. In the "100 µg + Alhydrogel" group, 13 out of 16 patient samples were analyzed due to 2 patients in the group withdrawing from the study and an insufficient serum sample from a third patient.
Measure: Geometric Mean (95% Confidence Interval); unit: Antibody Titer
Arm/Group | 2 µg + Alhydrogel | 10 µg + Alhydrogel | 30 µg + Alhydrogel | 100 µg + Alhydrogel
Number analyzed (Participants) | 6 | 6 | 15 | 13
Antibody Titer | 139.2 [19.0 to 1018] | 511.2 [79.5 to 3287] | 492.9 [202.4 to 1200] | 996.0 [510.0 to 1942]
Statistical Analysis 1: Comparison: 30 µg + Alhydrogel; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Significance of IgG values at study day 196 as compared to day 0 (pre-immune)
Statistical Analysis 2: Comparison: 100 µg + Alhydrogel; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Significance of IgG values at study day 196 as compared to day 0 (pre-immune)

5. Secondary Outcome: Assessment of Transmission Reducing Activity (TRA) of Malaria Parasite
Description: Assessment of TRA, as measured by the standard membrane feeding assay (SMFA), one month after the second vaccination (Study Day 84) in either the 30 μg or 100 μg dose groups.
Time Frame: 84 days
Measure: Mean (95% Confidence Interval); unit: % TRA
Arm/Group | 2 µg + Alhydrogel | 10 µg + Alhydrogel | 30 µg + Alhydrogel | 100 µg + Alhydrogel
Number analyzed (Participants) | 0 | 0 | 16 | 15
% TRA |  |  | 3.5 [-106.4 to 54.7] | 4.3 [-103.8 to 55.3]
Statistical Analysis 1: Comparison: 30 µg + Alhydrogel; Test type: Superiority or Other; p = 0.8, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 100 µg + Alhydrogel; Test type: Superiority or Other; p = 0.6, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Assessment of Transmission Reducing Activity (TRA) of Malaria Parasite
Description: Assessment of TRA, as measured by the standard membrane feeding assay (SMFA), showing ≥80% reduction of oocysts in Anopheles mosquito gut in ≥50% of the subjects with Study Day 196 sera (one month after the third vaccination) (Study Day 196) in either the 30 μg or 100 μg dose groups.
Time Frame: 196 days
Measure: Mean (95% Confidence Interval); unit: % TRA
Arm/Group | 2 µg + Alhydrogel | 10 µg + Alhydrogel | 30 µg + Alhydrogel | 100 µg + Alhydrogel
Number analyzed (Participants) | 0 | 0 | 15 | 13
% TRA |  |  | 9.1 [-92.1 to 56.9] | 22.5 [-59.8 to 62.9]
Statistical Analysis 1: Comparison: 30 µg + Alhydrogel; Test type: Superiority or Other; p = 0.5, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 100 µg + Alhydrogel; Test type: Superiority or Other; p = 0.3, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 7 months
Description: 196 days
Arm/Group | 2 µg + Alhydrogel | 10 µg + Alhydrogel | 30 µg + Alhydrogel | 100 µg + Alhydrogel
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 0/16 | 1/16
Other Adverse Events (participants affected / at risk) | 2/6 | 4/6 | 8/16 | 10/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 µg + Alhydrogel (N=6) | 10 µg + Alhydrogel (N=6) | 30 µg + Alhydrogel (N=16) | 100 µg + Alhydrogel (N=16)
Breast Abscess (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot Deformity (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2 µg + Alhydrogel (N=6) | 10 µg + Alhydrogel (N=6) | 30 µg + Alhydrogel (N=16) | 100 µg + Alhydrogel (N=16)
Fatigue/Malaise (General disorders) | 2 | 2 | 4 | 6
Headache (General disorders) | 0 | 3 | 5 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 5
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 3
Chills (General disorders) | 2 | 1 | 0 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Sweats (General disorders) | 0 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Fever (General disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In no event shall the PI publish or present, at any time, the data generated in the course of the performance of the study.